CLINICAL TRIAL: NCT05868135
Title: Guided Internet-delivered Treatment for Moderate Depression, Social Anxiety Disorder and Panic Disorder - An Open Naturalistic Multicentre Cost-effectiveness Trial
Brief Title: Effects and Cost-effectiveness of e-Meistring - a Guided Internet-delivered Psychological Treatment
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); The Hospital of Vestfold (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: 229387
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression Moderate; Anxiety, Social; Panic Disorder
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with moderate depression
  Interventions: Behavioral: eMeistring
- Patients with social anxiety disorder
  Interventions: Behavioral: eMeistring
- Patients with panic disorder
  Interventions: Behavioral: eMeistring

INTERVENTIONS:
Behavioral: eMeistring — Initial face-to-face visit, eight/nine sessions/modules of therapist guided ICBT, final face-to-face visit

SUMMARY:
The goal of this observational multicentre study is to address the effectiveness and cost-effectiveness of providing a therapist guided internet based cognitive behavioural therapy (ICBT) for common mental disorders in a routine healthcare setting.

Main research questions is 1) What is the effectiveness of guided internet based treatment for moderate depression, panic disorder and social anxiety disorder across clinics in routine care? 2) What is the cost-effectiveness of guided internet based treatment for moderate depression, panic disorder and social anxiety disorder across clinics? 3) Who benefits from guided internet-delivered treatment? 4) What are the predictors of drop-out from guided internet based treatment? 5) To what extent does user experiences of guided internet based treatment influence adherence and effectiveness? Participants will receive up to nine guided ICBT sessions (modules) and answer questionnaires covering symptoms severity, health related quality of life, work and social ability, user satisfaction and medication. All questionnaires are part of the standard patient follow up routines in the four treatment locations participating in the study. Analytical approach is to compare locations/clinics and subgroups of patients.

DETAILED DESCRIPTION:
The therapist guided internet based cognitive therapy (ICBT) cover moderate depression, social anxiety disorder (SAC) and panic disorder (PD).

The eMeistring-program is standard treatment in all four hospitals/locations participating in the study. Patients are recruited through the ordinary clinical patient pathways. After a pre-treatment assessment, an initial face-to-face visit takes place (T1). Patients are given the opportunity to participate in the study based on informed concent. Next, participants in the depression program will receive eight guided internet based cognitive behavioural therapy sessions or modules. Similarly SAC and PD patients will receive nine modules. Therapist guidance are provided at least once a week via a secure email system. When sessions are finished (T2), a new face-to-face visit with the therapist is offered.

Therapists are licensed health personnel e.g. psychologists, registered nurses and clinical social workers, working in the clinics.

Administrative data about covering organizational implementation of the eMeistring treatment program, personnel involved and level of treatment activity is collected separately.

Inclusion criteria's for eMeistring therapy: having moderate depression, panic disorder and social anxiety disorder as a primary disorder, and having computer and internet access.

Exclusion criteria: severe depression, suicidal impulses and thoughts, bipolar disorders, psychosis, substance abuse, unstable medication last month), severe reading or writing disabilities.

Adverse events are taken care of through routine follow-up according to the outpatient clinic responsibility. Any responses from patients indicating suicidal behaviour triggers email to the therapist with an urge to follow-up.

Planned statistical analyses include multivariate analyses of effectiveness (intention-to-treat and completers), predictor analyses of drop-out and adherence, and cost-effectiveness analyses based on health related quality of life, intervention costs and other health care and societal costs, analysing location specific differences stratified by patient groups.

ELIGIBILITY:
Inclusion Criteria:

Having moderate depression, panic disorder and social anxiety disorder as a primary disorder. Access to computer and internet.

Exclusion Criteria:

Having severe depression, suicidal impulses and thoughts, bipolar disorders, psychosis, substance abuse, unstable medication last month, severe reading or writing disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population living in the geographical areas in which provision of specialized health care services are the resonsibility of the four health enterprices/locations participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression severity | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For moderate depression group: Depression severity assessed by PHQ-9, Patient Health Questionnaire score. Minimum score is 0, maximum score is 27. Higher score indicates more severe depression
Social phobia | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For social anxiety group: Social Phobia assessed by SPIN, Social Phobia Inventory score. Minimum score is 0, maximum score is 68. Higher score indicates more severe phobia.
Panic disorder symptoms | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For panic disorder group: Panic disorder disorder symptoms assessed by PDSS-SR, Panic Disorder Severity Scale. Minimum raw score: 0, maximum raw score: 28. Composite scores range from 0-4. The composite score is the average of the seven items. Higher score indicates higher severity of panic disorder.

SECONDARY OUTCOMES:
Health Related Quality of Life | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For all patients: Health related quality of life assessed by EQ-5D-5L index score, EuroQol-5Dimension-5Level index score. Minimum score is 0, maximum score is 1. Higher score indicates higher health related quality of life.
Work and social adjustment | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For all patients: Work and social adjustment assessed by Work and Social Adjustment Scale score. Minimum score is 0, maximum score is 40. Higher score indicates worse level of social functioning.
Anxiety severity | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For all patients: Anxiety severity will be assessed by GAD-7, Generalized Anxiety Disorder 7-item score. Minimum score is 0, maximum score is 21. Higher score indicates more severe anxiety.
System Usability | Up to 14 weeks after treatment start (T2)
  For all patients: System usability will be assessed by the System Usability Scale Score. Minimum score is 0, maximum score is 100. Higher SUS scores indicate better usability.
Depression severity | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  For social anxiety group an panic disorder group: Depression severity assessed by PHQ-9, Patient Health Questionnaire score. Minimum score is 0, maximum score is 27. Higher score indicates more severe depression
Cost of health care services | Period between pre treatment (T1) and up to 14 weeks after treatment start (T2), and to six months after post treatment (T3) and until two years (T4)
  Cost of health care services calculated as sum costs for hospital inpatient stays plus outpatient visits plus home care visits plus nursing home stays plus general practitioner visits plus physiotherapist visits plus other supportive care visits.
Medication | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after T2 (T3) and after two years (T4)
  Patient reported use of medication, assessed by a separate questionnaire.
Work participation | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after post treatment (T3) and after two years (T4)
  Work participation assessed by questionnaire: Currently employed or not.
Sickness absenteeism | Pre treatment (T1), up to 14 weeks after treatment start (T2), six months after post treatment (T3) and after two years (T4)
  Sickness absenteeism assessed by questionnaire: Number of days absent the last four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Elin T Ulleberg, Master, Principal Investigator — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Helse Bergen HF, Bergen
  - Sykehuset Innlandet HF, Lillehammer
  - St. Olavs Hospital HF, Trondheim
  - Sykehuset i Vestfold HF, Tønsberg

IPD SHARING:
Plan to Share IPD: No